CLINICAL TRIAL: NCT01024192
Title: Efficacy and Safety Assessment of ZOlpidem (Stilnox CR) Administered on as Needed Basis in Patients With Chronic insomNIA
Brief Title: Efficacy and Safety Assessment of ZOlpidem (Stilnox CR) in Patients With Chronic insomNIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZOLPI_L_04134
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-10

CONDITIONS: Sleep Disorders
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Zolpidem

ARMS (1):
- 1 (Experimental): Zolpidem 12.5mg tablet at bed time during 12 weeks
  Interventions: Drug: ZOLPIDEM SL800750

INTERVENTIONS:
Drug: ZOLPIDEM SL800750 — Pharmaceutical form: Zopidem 12.5 mg tablets
  Route of administration: Oral
  Dose regimen:One tablet at bed time and as needed (the patients choose which night they take the tablet without limit of number of nights)

SUMMARY:
Primary Objective:

To evaluate the efficacy and safety of the use of Stilnox CR in Mexican patients with chronic insomnia at the prescription conditions of daily practice

Secondary Objective:

To evaluate the satisfaction of the patient with chronic insomnia with Stilnox CR over an as needed basis.

ELIGIBILITY:
Inclusion Criteria:

- Primary insomnia diagnosis (difficulty for initiating sleep, or maintaining sleep to wake up to early in the morning, or to present a restless sleep) which causes clinically significant disturbances in the areas of social, work functioning or other important areas

Exclusion criteria:

* Serious, severe and/or acute respiratory impairment
* Severe liver impairment
* Hypersensitivity to the formulation components or to some of its active metabolites
* Pregnant or breast-feeding women Patients with important associated disorders in SNC and specially psychotic disorders
* Patients with the probability of using alcoholic beverages concomitantly (as a precaution measure)
* Chronic use of benzodiazepines

Moreover, in order to follow the international regulations in terms of the use and handling of hypnotic compounds, and to guarantee the appropriate study performance, no patients with one or more of the following characteristics should be included:

* Patients who cannot comply to follow-up
* Patients who have any drug abuse problem
* Individuals who work changing night shifts or with pathological snoring
* Presence (or suspicion) of sleep apnea, periodical legs movements or restless legs syndrome

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2009-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Improvement of the Clinical Global Impression (CGI) score | At day 84 (visit 5)

SECONDARY OUTCOMES:
Illness severity and average change during the study | At day 1 (baseline), day 14 (visit 2), day 28 (visit 3), day 56 (visit 4) and day 84 (visit 5)
Pittsburgh Sleep Quality Index (PSQI) score | At day 1 (baseline), day 28 (visit 3), day 56 (visit 4) and day 84 (visit 5)
Patient satisfaction questionnaire | At day 84 (visit 5)
Safety evaluation via Adverse events reported | At day 14 (visit 2), day 28 (visit 3), day 56 (visit 4) and day 84 (visit 5)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Col. Coyoacan, Mexico